CLINICAL TRIAL: NCT03741790
Title: Airway Management of Pediatric Patients With Klippel-Feil Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Patcharee Sriswasdi, Attending staff, Boston Children's Hospital
Other Study IDs: IRB-P00029640
Record Dates: First submitted 2018-08-29; First posted 2018-11-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Klippel-Feil Syndrome
Keywords: airway; intubation
MeSH Terms: conditions — Klippel-Feil Syndrome | interventions — Ventilation; Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ventilation — The difficult mask ventilation is defined as A) It is not possible for unassisted anesthesiologist to maintain the SpO2 > 90% using 100% oxygen and positive pressure mask ventilation in a patient whose SpO2 > 90% before anesthetic intervention; and/or B) It is not possible for unassisted anesthesiologist to prevent or reverse signs of inadequate ventilation during positive mask ventilation.
Procedure: Intubation — The difficult endotracheal intubation is defined as " It is not possible to visualize any portion of the vocal cords with conventional laryngoscopy" or when proper insertion of the endotracheal tube with conventional laryngoscopy requires more than three attempts or more than ten minutes.

SUMMARY:
Klippel-Feil syndrome (KFS) was first described in 1912 by Klippel and Feil as a classic triad are comprised of a short neck, a low posterior hairline and restricted motion of the neck. This disease is considered as one of the congenital causes of difficult airway with the incidence of 1:42,000 live births.

The current research findings suggested that the difficulties of airway management for KFS increases with age. In pediatric patients, the airway of those patients can be managed without difficulties. For adults, the fiberoptic-assisted intubation is also suggested.

The purpose of this study is to review the airway management of pediatric patients with KFS to provide recommendation of airway management for these patients. A retrospective electronic chart review will be conducted by using Boston Children's Hospital (BCH) database, which identified patients with KFS who had undergone general anesthesia from June 2012 to June 2018.

DETAILED DESCRIPTION:
Klippel-Feil syndrome (KFS) was first described in 1912 by Klippel and Feil as a classic triad are comprised of a short neck, a low posterior hairline and restricted motion of the neck due to fused cervical vertebrae with the incidence of 1:42,000 live births1,2. The etiology is presumed to involve in PAX gene family mutation defect and Notch signaling pathway. KFS patients are classified into 3 types based on the location of fusion; Type 1 patients have a single congenitally fused cervical segment; Type 2 patients show multiple non-contiguous, congenitally fused cervical segments; and Type 3 patients show multiple contiguous, congenitally fused cervical segments. In 1974, Hensinger et al studied 50 KFS patients aged 4 to 34 years and their associated anomalies. The findings revealed less than half had the classic triad of findings, more than half had scoliosis and a third had renal anomalies. All patients were at risk of having other serious anomalies such as Sprengel's deformity, hearing impairment, synkinesia and congenital heart disease.

The current literature focused on isolated case reports suggested an awake fiberoptic intubation as a safest option to secure airway in adult patient with KFS. For pediatric patients with KFS, their airway management could be challenging, there is no literature report describing unsuccessful or difficult mask ventilation or LMA insertion. Bakan et al reported an overview of direct laryngoscopy for tracheal intubation in KFS patients aged 26 days to 16 years old, 18 of 25 cases were successfully intubated by direct laryngoscope (DL). From 13 literatures reviewed by Bakan et al, there is no report of an unsuccessful DL in children with KFS younger than 4 years. Despite the formidable appearance for airway management, recent pediatric data encourage the anesthesia providers to perform DL instead of fiberoptic intubation. However, a successful DL event in anesthesia history record does not guarantee an ease of next DL event because the airway of KFS patients are progressively worse over time.

The investigators propose a retrospective electronic chart review of patients with KFS who had undergone general anesthesia in Boston Children's Hospital from June 2012 to June 2018. The purpose of this study is to review the airway management techniques of pediatric patients with KFS and provide recommendation of airway management for these patients. A retrospective electronic chart review will be conducted by using Boston Children's Hospital (BCH) database, which identified patients with KFS who had undergone general anesthesia from June 2012 to June 2018.

The investigators hope to provide specific anatomical abnormalities and age of pediatric patients with KFS to suggest they are at risk of difficult airway. Finally, the investigators hope this information can be used to suggest a proper choice of airway management for specific type and age group of KFS patients.

ELIGIBILITY:
Inclusion Criteria:

* All KFS patients who scheduled for surgery at BCH from June 2012 to June 2018.

Exclusion Criteria:

* Patients with incomplete or absent of medical records on AIMS such as ventilation and intubation technique are not clearly document.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All KFS patients who scheduled for surgery at BCH from June 2012 to June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of difficult airway cases among KFS is defined by using the ASA task force definition. | We will collect data on a day of surgery from patient's arrival into their induction and intubation period, and through their postoperative period upto 1 week.
  The difficult airway is defined as "The clinical situation in which a conventionally trained anesthesiologist experiences difficulty with mask ventilation, difficulty with tracheal intubation, or both".

SECONDARY OUTCOMES:
Specific anatomical abnormalities of KFS patients which related to difficult airway | We will collect data on a day of surgery from patient's arrival into their induction and intubation period, and through their postoperative period upto 1 week
  Specific anatomical abnormalities of KFS patients who had difficult airway is define by radiological classification based on the location of fusion; Type 1 patients have a single congenitally fused cervical segment; Type 2 patients show multiple non-contiguous, congenitally fused cervical segments; and Type 3 patients show multiple contiguous, congenitally fused cervical segments.

CONTACTS AND LOCATIONS:
Overall Officials: Patcharee Sriswasdi, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston children's hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We might share individual participant data if it allows maximum use of the data.

REFERENCES:
- [Background] Hase Y, Kamekura N, Fujisawa T, Fukushima K. Repeated anesthetic management for a patient with Klippel-Feil syndrome. Anesth Prog. 2014 Fall;61(3):103-6. doi: 10.2344/0003-3006-61.3.103. PMID 25191983
- [Background] Altay N, Yuce HH, Aydogan H, Dorterler ME. Airway management in newborn with Klippel-Feil syndrome. Braz J Anesthesiol. 2016 Sep-Oct;66(5):551-3. doi: 10.1016/j.bjane.2014.03.006. Epub 2014 Apr 29. PMID 27591474
- [Background] Stallmer ML, Vanaharam V, Mashour GA. Congenital cervical spine fusion and airway management: a case series of Klippel-Feil syndrome. J Clin Anesth. 2008 Sep;20(6):447-51. doi: 10.1016/j.jclinane.2008.04.009. PMID 18929286
- [Background] Raj D, Luginbuehl I. Managing the difficult airway in the syndromic child. Continuing Education in Anaesthesia Critical Care & Pain. 2015;15(1):7-13.
- [Background] Khawaja OM, Reed JT, Shaefi S, Chitilian HV, Sandberg WS. Crisis resource management of the airway in a patient with Klippel-Feil syndrome, congenital deafness, and aortic dissection. Anesth Analg. 2009 Apr;108(4):1220-5. doi: 10.1213/ane.0b013e3181957d9b. PMID 19299791
- [Background] Samartzis DD, Herman J, Lubicky JP, Shen FH. Classification of congenitally fused cervical patterns in Klippel-Feil patients: epidemiology and role in the development of cervical spine-related symptoms. Spine (Phila Pa 1976). 2006 Oct 1;31(21):E798-804. doi: 10.1097/01.brs.0000239222.36505.46. PMID 17023841
- [Background] Hensinger RN, Lang JE, MacEwen GD. Klippel-Feil syndrome; a constellation of associated anomalies. J Bone Joint Surg Am. 1974 Sep;56(6):1246-53. PMID 4436358
- [Background] Bakan M, Umutoglu T, Zengin SU, Topuz U. The success of direct laryngoscopy in children with Klippel-Feil Syndrome. Minerva Anestesiol. 2015 Dec;81(12):1384-6. Epub 2015 Sep 18. No abstract available. PMID 26381356